CLINICAL TRIAL: NCT00258167
Title: Family Involvement in The Treatment Of a Mentally Ill Relative
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lev-Hasharon Mental Healtlh Center (Other Government)
Responsible Party: Dr. Igor Oyffe, Lev Hasharon Mental Health Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: LH12/2005.CTIL
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Families of Mentally Ill
Keywords: Family members; Illness burden; Mental Disorders; Family intervention
MeSH Terms: conditions — Mental Disorders

INTERVENTIONS:
Behavioral: filling the "Experience of Caregiving Inventory" — 8 weeks of group therapy for family members

SUMMARY:
* Research demonstrates that the families of the seriously mentally ill are burdened by this caregiving role and by their responsibilities
* Research also demonstrates that family interventions are effective and that they have a potential to reduce family burden, as well as to improve the condition of the mentally ill patients.
* We assume that the sibling group intervention would be effective in reducing the family burden of the siblings, and that this reduction would be reflected in their replies to the "Experience of Caregiving Inventory".

DETAILED DESCRIPTION:
* The group for siblings is an intervention which is carried out in the outpatient clinic of Lev HaSharon Mental Health Center in cycles which last eight weeks;
* Every group cycle will include between 10-14 participants, all siblings of persons with mental illness. The patients themselves (ill siblings) are either hospitalized in Lev HaSharon Mental Health Center, or are outpatients in the Lev HaSharon Mental Health Outpatient Unit, or in the community at large.
* The group is an ongoing group: short term intensive group intervention in a dynamic orientation. Veteran participants of each cycle are welcome to re-join at following cycles, and at the same time new participants can join at the beginning of each cycle.
* Participants will be asked to fill the "Experience of Caregiving Inventory" twice: first time before the first meeting of a particular cycle of sibling group and second time: after the last (eighth) meeting of this group cycle.

ELIGIBILITY:
Inclusion Criteria:

* siblings of persons with mental illness

Exclusion Criteria:

* persons junior then 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-11; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Score on the "Experience of Caregiving Inventory" following 8 weeks of participation in the group. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Igor Oyffe, MD, Principal Investigator — Lev-Hasharon Mental Healtlh Center
Locations (1):
- Lev-HasharonMHC, Netanya, Israel

REFERENCES:
- [Background] Melamed, S. Permission: A conceptual tool for treating mentally ill patients and their families. Journal of Family Psychotherapy. 12 (2). Pp. 29-42, 2001.
- [Background] Dixon L, McFarlane WR, Lefley H, Lucksted A, Cohen M, Falloon I, Mueser K, Miklowitz D, Solomon P, Sondheimer D. Evidence-based practices for services to families of people with psychiatric disabilities. Psychiatr Serv. 2001 Jul;52(7):903-10. doi: 10.1176/appi.ps.52.7.903. PMID 11433107